CLINICAL TRIAL: NCT04634877
Title: A Phase 3, Randomized, Double-Blind Study of Pembrolizumab Versus Placebo in Combination With Adjuvant Chemotherapy With or Without Radiotherapy for the Treatment of Newly Diagnosed High-Risk Endometrial Cancer After Surgery With Curative Intent (KEYNOTE-B21 / ENGOT-en11 / GOG-3053)
Brief Title: Study of Pembrolizumab (MK-3475) in Combination With Adjuvant Chemotherapy With or Without Radiotherapy in Participants With Newly Diagnosed Endometrial Cancer After Surgery With Curative Intent (MK-3475-B21 / KEYNOTE-B21 / ENGOT-en11 / GOG-3053)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: European Network for Gynaecological Oncological Trial Groups (Unknown); Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-B21; KEYNOTE-B21 (Other: MSD); ENGOT-en11 (Other: European Network for Gynaecological Oncological Trial groups); GOG-3053 (Other: Gynecologic Oncology Group); jRCT2031200399 (Registry Identifier: jRCT); 2022-501973-37-00 (Registry Identifier: EU CT); U1111-1282-6430 (Registry Identifier: UTN); 2020-003424-17 (EudraCT Number)
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2025-06-09 (Actual); Status verified 2025-05

CONDITIONS: Endometrial Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2 )
MeSH Terms: conditions — Endometrial Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Carboplatin; Paclitaxel; Docetaxel; Cisplatin; Brachytherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Chemotherapy (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for 6 cycles followed by pembrolizumab 400 mg IV on Day 1 of each 6-week cycle (Q6W) for an additional 6 cycles. During the Q3W dosing period of pembrolizumab, participants receive concurrent standard of care (SoC) chemotherapy for 4 or 6 cycles. Participants optionally receive radiotherapy starting within 6 weeks of completion of SoC chemotherapy. The SoC chemotherapy regimen includes carboplatin AUC 5 or 6 IV Q3W plus paclitaxel 175 mg/m^2 IV Q3W. In the event of severe hypersensitivity to, or an AE requiring discontinuation of, carboplatin or paclitaxel, cisplatin or docetaxel may be substituted after investigator consults with sponsor. The SoC radiotherapy regimen may include, at the discretion of the investigator, external beam radiotherapy (EBRT) ≥4500 cGY with variable dose frequency, with or without cisplatin 50 mg/m^2 IV on days 1 and 29 of EBRT, and/or brachytherapy radiation.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Docetaxel; Drug: Cisplatin; Radiation: External Beam Radiotherapy (EBRT); Drug: Cisplatin (as radiosensitizer); Radiation: Brachytherapy
- Placebo + Chemotherapy (Placebo Comparator): Participants receive placebo to pembrolizumab intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for 6 cycles followed by placebo IV on Day 1 of each 6-week cycle (Q6W) for an additional 6 cycles. During the Q3W dosing period of placebo, participants receive concurrent standard of care (SoC) chemotherapy for 4 or 6 cycles. Participants optionally receive radiotherapy starting within 6 weeks of completion of SoC chemotherapy. The SoC chemotherapy regimen includes carboplatin AUC 5 or 6 IV Q3W plus paclitaxel 175 mg/m^2 IV Q3W. In the event of severe hypersensitivity to, or an AE requiring discontinuation of, carboplatin or paclitaxel, cisplatin or docetaxel may be substituted after investigator consults with sponsor. The SoC radiotherapy regimen may include, at the discretion of the investigator, external beam radiotherapy (EBRT) ≥4500 cGY with variable dose frequency, with or without cisplatin 50 mg/m^2 IV on days 1 and 29 of EBRT, and/or brachytherapy radiation.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Placebo for pembrolizumab; Drug: Docetaxel; Drug: Cisplatin; Radiation: External Beam Radiotherapy (EBRT); Drug: Cisplatin (as radiosensitizer); Radiation: Brachytherapy

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab + Chemotherapy
Drug: Carboplatin — IV infusion
Drug: Paclitaxel — IV infusion
Drug: Placebo for pembrolizumab — IV infusion
  Arms: Placebo + Chemotherapy
Drug: Docetaxel — IV infusion docetaxel 75 mg/m^2 Q3W or 25 mg/m2 QW may be given in place of paclitaxel following sponsor consultation if a participant experiences severe hypersensitivity to paclitaxel or an adverse event requiring discontinuation of paclitaxel.
Drug: Cisplatin — Cisplatin 75 mg/m^2 IV infusion Q3W may be given in place of carboplatin following sponsor consultation if a participant experiences severe hypersensitivity to carboplatin or an adverse event requiring discontinuation of carboplatin.
  Other Names: Platinol®; Platinol®-AQ
Radiation: External Beam Radiotherapy (EBRT) — ≥4500 cGY given according to local practice, at the discretion of the investigator
Drug: Cisplatin (as radiosensitizer) — If a participant receives external beam radiotherapy (EBRT), then cisplatin 50 mg/m^2 IV infusion may be administered as a radiosensitizer at the discretion of the investigator, on days 1 and 29
  Other Names: Platinol®; Platinol®-AQ
Radiation: Brachytherapy — Given according to local practice, at the discretion of the investigator
  Other Names: Internal radiation therapy

SUMMARY:
The purpose of this study is to compare pembrolizumab + adjuvant chemotherapy with placebo + adjuvant chemotherapy, with or without radiotherapy, with respect to disease-free survival (DFS) as assessed radiographically by the investigator or by histopathologic confirmation of suspected disease recurrence, and with respect to overall survival (OS). The primary hypotheses are that pembrolizumab + adjuvant chemotherapy is superior to placebo + adjuvant chemotherapy, with or without radiotherapy, with respect to DFS as assessed radiographically by the investigator or by histopathologic confirmation of suspected disease recurrence, and with respect to OS.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed new diagnosis of Endometrial Carcinoma or Carcinosarcoma (Mixed Mullerian Tumor) and:

  * Has undergone curative intent surgery that included hysterectomy and bilateral salpingo-oophorectomy; and
  * Is at high risk for recurrence following treatment with curative intent surgery, ie: Fédération Internationale de Gynécologie et d'Obstétrique (FIGO) 2009 surgical stage I/II with myometrial invasion of non-endometrioid histology; FIGO 2009 surgical stage I/II with myometrial invasion of any histology with known aberrant p53 expression or p53 mutation; or FIGO (2009) surgical stage III or IVA of any histology.
* Is disease-free with no evidence of loco-regional disease or distant metastasis post operatively and on imaging.
* Has not received any radiation or systemic therapy, including immunotherapy, hormonal therapy, or hyperthermic intraperitoneal chemotherapy (HIPEC), in any setting including the neoadjuvant setting for endometrial cancer (EC).
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days before randomization.
* Submission of a tumor tissue sample from current diagnosis of Endometrial Carcinoma or Carcinosarcoma for prospective determination of histology and mismatch repair (MMR) status by central vendor is required for all participants.
* Has adequate organ function within 7 days of randomization.

Exclusion Criteria:

* Has recurrent endometrial carcinoma or carcinosarcoma.
* Has uterine mesenchymal tumor such as an endometrial stromal sarcoma, leiomyosarcoma, or other types of pure sarcomas. Adenosarcomas are also not allowed.
* Has FIGO (2009) Surgical Stage I/II EC of endometrioid histology without a known aberrant p53 expression or p53 mutation.
* Is known to have a deoxyribonucleic acid (DNA) polymerase epsilon catalytic subunit A (POLE) mutation.
* Has FIGO Stage IVB disease of any histology even if there is no evidence of disease after surgery.
* Has residual tumor whether measurable or non-measurable after surgery.
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 3 years.

  * Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in situ cancers.
* Has received prior therapy with an anti-programmed cell death receptor 1 (PD-1), anti-programmed cell death receptor ligand 1 (PD-L1), or anti-programmed cell death receptor ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137).
* Has received a live vaccine within 30 days before the first dose of study intervention.

  * Note: killed vaccines are allowed.
* Has a known intolerance to study intervention (or any of the excipients).
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention.

  * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has any contraindication to the use of carboplatin or paclitaxel.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of HIV infection.
* Has a known history of Hepatitis B or known active Hepatitis C virus infection.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Has had an allogenic tissue/solid organ transplant.
* Has not recovered adequately from surgery and/or any complications from the surgery.
* Is breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) as Assessed Radiographically by Investigator or by Histopathologic Confirmation of Suspected Disease Recurrence | Up to approximately 42 months
  DFS is defined as the time from randomization to the first documented local recurrence, distant metastasis, secondary systemic malignancy, or death due to any cause, whichever occurs first. The DFS as assessed radiographically by investigator or by histopathologic confirmation of suspected disease recurrence, will be presented.
Overall Survival (OS) | Up to approximately 54 months
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) as Assessed Radiographically by Blinded Independent Central Review (BICR) or by Histopathologic Confirmation of Suspected Disease Recurrence | Up to approximately 42 months
  DFS is defined as the time from randomization to the first documented local recurrence, distant metastasis, secondary systemic malignancy, or death due to any cause, whichever occurs first. The DFS as assessed radiographically by BICR or by histopathologic confirmation of suspected disease recurrence, will be presented.
Disease-Free Survival (DFS) as Assessed Radiographically by Investigator or by Histopathologic Confirmation of Suspected Disease Recurrence by Combined Positivity Score (CPS)-Determined Programmed Cell Death 1 Ligand 1 (PD-L1) Status | Up to approximately 42 months
  DFS is defined as the time from randomization to the first documented local recurrence, distant metastasis, secondary systemic malignancy, or death due to any cause, whichever occurs first. The DFS as assessed radiographically by investigator or by histopathologic confirmation of suspected disease recurrence by CPS-determined PD-L1 status will be presented.
Overall Survival (OS) as Assessed Radiographically by Investigator or by Histopathologic Confirmation of Suspected Disease Recurrence by Combined Positivity Score (CPS)-Determined Programmed Cell Death 1 Ligand 1 (PD-L1) Status | Up to approximately 54 months
  OS is defined as the time from randomization to death due to any cause. The OS as assessed radiographically by investigator or by histopathologic confirmation of suspected disease recurrence by CPS-determined PD-L1 status will be presented.
Disease-Free Survival (DFS) as Assessed Radiographically by Investigator or by Histopathologic Confirmation of Suspected Disease Recurrence by Tumor Mutation Burden (TMB) Status | Up to approximately 42 months
  DFS is defined as the time from randomization to the first documented local recurrence, distant metastasis, secondary systemic malignancy, or death due to any cause, whichever occurs first. The DFS as assessed radiographically by investigator or by histopathologic confirmation of suspected disease recurrence by tumor mutation burden (TMB) status, will be presented.
Overall Survival (OS) as Assessed Radiographically by Investigator or by Histopathologic Confirmation of Suspected Disease Recurrence by Tumor Mutation Burden (TMB) Status | Up to approximately 54 months
  OS is defined as the time from randomization to death due to any cause. The OS as assessed radiographically by investigator or by histopathologic confirmation of suspected disease recurrence by tumor mutation burden (TMB) status will be presented.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 54 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to approximately 52 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be presented.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Global Health Status/Quality of Life (QoL) Score | Baseline and up to approximately 54 months
  The EORTC QLQ-C30 is a questionnaire that rates the overall quality of life in cancer participants. Participant responses to questions 29 ("How would you rate your overall health during the past week?") and 30 ("How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). A higher score indicates a better overall health/quality of life status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined scores will be presented.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Physical Function Score | Baseline and up to approximately 54 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=not at all to 4=very much). A higher score indicates a better quality of life. The change from baseline in physical function (EORTC QLQ-C30 Items 1-5) score will be presented.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Symptom Specific Scale for Endometrial Cancer (EORTC QLQ-EN24) Score | Baseline and up to approximately 54 months
  The EORTC-QLQ-EN24 is a 24-item questionnaire developed to be used in conjunction with the EORTC-QLQ-C30 to assess the quality of life of endometrial cancer patients. Participant responses are scored on a 4-point scale (1=not at all to 4=very much). A higher score indicates a better quality of life. The change from baseline in EORTC QLQ-E24 score will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (231):
- United States (29):
  - University of Alabama - Birmingham ( Site 3061), Birmingham, Alabama
  - University of South Alabama, Mitchell Cancer Institute ( Site 3058), Mobile, Alabama
  - HonorHealth Research Institute - Biltmore ( Site 3043), Phoenix, Arizona
  - Arizona Oncology Associates PC- HOPE ( Site 3049), Tucson, Arizona
  - UCSD Moores Cancer Center ( Site 3053), La Jolla, California
  - University Of Colorado ( Site 3051), Aurora, Colorado
  - Smilow Cancer Hospital at Yale New Haven ( Site 3070), New Haven, Connecticut
  - Mount Sinai Cancer Center ( Site 3081), Miami Beach, Florida
  - Northside Hospital ( Site 3036), Atlanta, Georgia
  - Northwestern Memorial Hospital ( Site 3044), Chicago, Illinois
  - Parkview Cancer Institute ( Site 3067), Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center ( Site 3071), Indianapolis, Indiana
  - University of Iowa Hospital and Clinics ( Site 3046), Iowa City, Iowa
  - Norton Cancer Institute - St. Matthews ( Site 3056), Louisville, Kentucky
  - WK Physicians Network/Gynecologic Oncology Associates ( Site 3047), Shreveport, Louisiana
  - University of Massachusetts Medical School ( Site 3037), Worcester, Massachusetts
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 3076), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 3042), New York, New York
  - Montefiore Medical Center ( Site 3065), The Bronx, New York
  - Duke Cancer Center ( Site 3072), Durham, North Carolina
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 3080), Fargo, North Dakota
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive C, Columbus, Ohio
  - Legacy Good Samaritan Medical Center ( Site 3033), Portland, Oregon
  - Sidney Kimmel Cancer Center - Jefferson Health ( Site 3078), Philadelphia, Pennsylvania
  - AHN West Penn Hospital ( Site 3060), Pittsburgh, Pennsylvania
  - Abington Hospital - Asplundh Cancer Center ( Site 3073), Willow Grove, Pennsylvania
  - Sanford Gynecology Oncology ( Site 3045), Sioux Falls, South Dakota
  - UT Southwestern Medical Center ( Site 3063), Dallas, Texas
  - VCU Massey Cancer Center ( Site 3068), Richmond, Virginia
- Argentina (9):
  - Centro de Oncología e Investigación de Buenos Aires ( Site 1005), Berazategui, Buenos Aires
  - IDIM Instituto de Diagnostico e Investigaciones Metabolicas ( Site 1006), Caba, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 1003), Mar del Plata, Buenos Aires
  - Hospital Britanico de Buenos Aires ( Site 1002), Buenos Aires, Buenos Aires F.D.
  - Instituto de Oncologia de Rosario ( Site 1004), Rosario, Santa Fe Province
  - IDIM - Instituto de Diagnóstico e Investigaciones Metabólicas ( Site 1010), Buenos Aires
  - Hospital Aleman ( Site 1001), Buenos Aires
  - CEMIC ( Site 1009), Buenos Aires
  - Centro Oncologico Riojano Integral ( Site 1007), La Rioja
- Austria (2):
  - Medizinische Universitat Graz ( Site 2004), Graz, Styria
  - Medizinische Universitaet Innsbruck ( Site 2001), Innsbruck, Tyrol
- Belgium (11):
  - Saint-Luc UCL ( Site 2042), Brussels, Bruxelles-Capitale, Region de
  - C.I.U. Hopital Ambroise Pare ( Site 2039), Mons, Hainaut
  - CHR Verviers ( Site 2035), Verviers, Liege
  - OLV Ziekenhuis ( Site 2038), Aalst, Oost-Vlaanderen
  - AZ Maria Middelares Gent ( Site 2032), Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Gent ( Site 2037), Ghent, Oost-Vlaanderen
  - AZ Nikolaas ( Site 2031), Sint-Niklaas, Oost-Vlaanderen
  - UZ Leuven ( Site 2040), Leuven, Vlaams-Brabant
  - AZ Groeninge ( Site 2036), Kortrijk, West-Vlaanderen
  - CHC - Groupe Sante ( Site 2041), Liège
  - CHU Liege Sart-Tilman ( Site 2044), Liège
- Canada (5):
  - Tom Baker Cancer Centre ( Site 3007), Calgary, Alberta
  - Kingston Health Sciences Centre ( Site 3003), Kingston, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 3006), Montreal, Quebec
  - McGill University Health Centre ( Site 3005), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 3, Québec, Quebec
- Chile (5):
  - Fundacion Arturo Lopez Perez FALP ( Site 1062), Santiago, Region M. de Santiago
  - Centro de Cancer Nuestra Senora de la Esperanza ( Site 1063), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 1070), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 1061), Temuco, Región de la Araucanía
  - Oncocentro ( Site 1065), Viña del Mar, Región de Valparaíso
- China (24):
  - Anhui Provincial Hospital-Obstetrics and Gynecology ( Site 4034), Hefei, Anhui
  - Beijing Cancer Hospital ( Site 4048), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 4036), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 4040), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University ( Site 4060), Xiamen, Fujian
  - The First Affiliated Hospital ( Site 4043), Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 4049), Nanning, Guangxi
  - Harbin Medical University Cancer Hospital ( Site 4033), Harbin, Heilongjiang
  - Hubei Cancer Hospital ( Site 4059), Wuhan, Hubei
  - Xiangya Hospital Central-South University ( Site 4035), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 4050), Changsha, Hunan
  - Nanjing Drum Tower Hospital ( Site 4037), Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital ( Site 4051), Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University ( Site 4057), Changchun, Jilin
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 4045), Xi'an, Shaanxi
  - Obstetrics and Gynecology Hosp. Fudan University ( Site 4041), Shanghai, Shanghai Municipality
  - Shanghai Renji Hospital Affiliated to Jiao Tong University ( Site 4053), Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital-Gynecology department ( Site 4001), Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital ( Site 4039), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital ( Site 4054), Tianjin, Tianjin Municipality
  - Yunnan Province Cancer Hospital-Gynecology Department ( Site 4055), Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University-Gynecology ( Site 4002), Hangzhou, Zhejiang
  - Women s Hospital School of Medicine Zhejiang University ( Site 4032), Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 4056), Wenzhou, Zhejiang
- Colombia (4):
  - Clínica Vida Fundación - Sede Poblado ( Site 1096), Medellín, Antioquia
  - Instituto Nacional de Cancerología E.S.E ( Site 1094), Bogotá, Bogota D.C.
  - Instituto Cancerologico de Narino Ltda ( Site 1092), Pasto, Departamento de Nariño
  - Fundacion Valle del Lili ( Site 1093), Cali, Valle del Cauca Department
- Czechia (4):
  - Fakultní nemocnice Brno Bohunice-Gynekologicko-porodnicka klinika ( Site 2394), Brno, Brno-mesto
  - Fakultni nemocnice Kralovske Vinohrady ( Site 2393), Prague, Praha 10
  - Vseobecna fakultni nemocnice v Praze ( Site 2391), Prague, Praha 2
  - Fakultni nemocnice Olomouc ( Site 2392), Olomouc
- Denmark (5):
  - Rigshospitalet University Hospital ( Site 2515), Copehagen, Capital Region
  - Herlev Hospital ( Site 2514), Herlev, Capital Region
  - Aalborg Universitetshospital ( Site 2511), Aalborg, North Denmark
  - Roskilde Sygehus ( Site 2513), Roskilde, Region Sjælland
  - Odense Universitetshospital ( Site 2512), Odense, Region Syddanmark
- Finland (3):
  - Kuopio University Hospital ( Site 2543), Kuopio, Northern Savonia
  - Tampere University Hospital ( Site 2541), Tampere, Pirkanmaa
  - Turku University Hospital ( Site 2542), Turku, Southwest Finland
- France (12):
  - Institut De Cancerologie De Lorraine ( Site 2072), Vandœuvre-lès-Nancy, Ain
  - Centre Antoine Lacassagne ( Site 2073), Nice, Alpes-Maritimes
  - Centre Francois Baclesse ( Site 2062), Caen, Calvados
  - Hôpital Privé Des Côtes d'Armor ( Site 2063), Plérin, Cotes-d Armor
  - CHU Besancon - Hopital Jean Minjoz ( Site 2068), Besançon, Doubs
  - Institut Bergonie ( Site 2067), Bordeaux, Gironde
  - Institut Universitaire du Cancer Toulouse - Oncopole ( Site 2065), Toulouse, Haute-Garonne
  - Institut Regional du Cancer de Montpellier - ICM ( Site 2069), Montpellier, Herault
  - Hopital prive du Confluent ( Site 2061), Nantes, Loire-Atlantique
  - Centre Hospitalier Lyon Sud ( Site 2064), Pierre-Bénite, Rhone
  - Hopital Cochin ( Site 2070), Paris, Île-de-France Region
  - Gustave Roussy ( Site 2071), Villejuif, Île-de-France Region
- Germany (8):
  - SLK-Kliniken Heilbronn GmbH ( Site 2116), Heilbronn, Baden-Wurttemberg
  - Klinikum Ludwigsburg ( Site 2111), Ludwigsburg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen ( Site 2113), Tübingen, Baden-Wurttemberg
  - Medizinische Hochschule Hannover-Department of Obstetrics and Gynecology ( Site 2109), Hanover, Lower Saxony
  - Universitätsklinikum Bonn-Gynaecological oncology ( Site 2103), Bonn, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung ( Site 2105), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Frauenheilkunde und Gebur, Dresden, Saxony
  - Universitätsklinikum Schleswig-Holstein ( Site 2101), Lübeck, Schleswig-Holstein
- Greece (6):
  - General Hospital of Patras. St Andrews ( Site 2421), Pátrai, Achaia
  - Geniko Panepistimako Nosokomeio ARETEIO ( Site 2423), Athens, Attica
  - Perifereiako Geniko Nosokomeio ALEXANDRA ( Site 2425), Athens, Attica
  - Athens University Hospital ATTIKON ( Site 2424), Chaïdári, Attica
  - Hospital Hygeia ( Site 2426), Marousi, Attica
  - Euromedica General Clinic of Thessaloniki ( Site 2422), Thessaloniki
- Israel (5):
  - Rambam Medical Center ( Site 2307), Haifa
  - Edith Wolfson Medical Center ( Site 2306), Holon
  - Hadassah Medical Center. Ein Kerem ( Site 2303), Jerusalem
  - Rabin Medical Center ( Site 2305), Petah Tikva
  - Chaim Sheba Medical Center ( Site 2301), Ramat Gan
- Italy (10):
  - Istittuto Nazionale dei Tumori Regina Elena IRCCS - IFO ( Site 2121), Roma, Abruzzo
  - Fondazione Policlinico Universitario Agostino Gemelli ( Site 2124), Rome, Lazio
  - Istituto di Candiolo - IRCCS ( Site 2125), Candiolo, Piedmont
  - Azienda Ospedaliera Spedali Civili di Brescia ( Site 2135), Brescia
  - IRCCS Ospedale San Raffaele ( Site 2130), Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 2122), Milan
  - Istituto Europeo di Oncologia IRCCS-Divisione di Ginecologia Oncologica ( Site 2132), Milan
  - Azienda Ospedaliera Universitaria Federico II ( Site 2123), Napoli
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 2127), Napoli
  - Istituto Oncologico Veneto IRCCS-Oncologia 2 ( Site 2134), Padua
- Japan (17):
  - Aichi Cancer Center Hospital ( Site 4190), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 4197), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 4181), Matsuyama, Ehime
  - Ehime University Hospital ( Site 4187), Tōon, Ehime
  - Kurume University Hospital ( Site 4186), Kurume, Fukuoka
  - Gunma Prefectural Cancer Center ( Site 4183), Ōta, Gunma
  - Hokkaido University Hospital ( Site 4194), Sapporo, Hokkaido
  - Hyogo Cancer Center ( Site 4195), Akashi, Hyōgo
  - Iwate Medical University Hospital ( Site 4189), Shiwa-gun, Iwate
  - University of the Ryukyus Hospital ( Site 4184), Nakagami-gun, Okinawa
  - Saitama Medical University International Medical Center ( Site 4182), Hidaka, Saitama
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 4192), Sunto-gun, Shizuoka
  - National Hospital Organization Kyushu Cancer Center ( Site 4193), Fukuoka
  - Niigata Cancer Center Hospital ( Site 4185), Niigata
  - Osaka International Cancer Institute ( Site 4188), Osaka
  - The Cancer Institute Hospital of JFCR ( Site 4196), Tokyo
  - Keio University Hospital ( Site 4191), Tokyo
- Mexico (7):
  - Investigacion Onco Farmaceutica S de RL de CV ( Site 1127), La Paz, Baja California Sur
  - Hospital San Lucas Cardiologica del Sureste ( Site 1122), Tuxtla Gutiérrez, Chiapas
  - Instituto Nacional de Cancerologia ( Site 1124), Mexico City, Mexico City
  - Christus Muguerza Clinica Vidriera ( Site 1125), Monterrey, Nuevo León
  - I Can Oncology Center SA de CV ( Site 1126), Monterrey, Nuevo León
  - Centro Oncologico Internacional. SEDNA ( Site 1121), Mexico City
  - Hospital Angeles Roma ( Site 1123), Mexico City
- Norway (3):
  - University Hospital of North Norway ( Site 2153), Tromsø, Troms
  - Soerlandet sykehus HF Kristiansand ( Site 2152), Kristiansand, Vest-Agder
  - Oslo Universitetssykehus Radiumhospitalet ( Site 2151), Oslo
- Poland (7):
  - Wielkopolskie Centrum Onkologii im.M.Sklodowskiej-Curie ( Site 2484), Poznan, Greater Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 2487), Siedlce, Masovian Voivodeship
  - Szpital Kliniczny im Ks Anny Mazowieckiej ( Site 2481), Warsaw, Masovian Voivodeship
  - Bialostockie Centrum Onkologii ( Site 2483), Bialystok, Podlaskie Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 2482), Gliwice, Silesian Voivodeship
  - SPZOZ MSWIA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie ( Site 2486), Olsztyn, Warmian-Masurian Voivodeship
  - Swietokrzyskie Centrum Onkologii SPZOZ ( Site 2485), Kielce, Świętokrzyskie Voivodeship
- Russia (13):
  - Arkhangelsk Clinical Oncological Dispensary ( Site 2637), Arkhangelsk, Arkhangelskaya oblast
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 2645), Ufa, Baskortostan, Respublika
  - Chelyabinsk Regional Clinical Center Oncology and Nuclear Medicine ( Site 2644), Chelyabinsk, Chelyabinsk Oblast
  - Krasnoyarsk Regional Clinical oncology dispensary ( Site 2643), Krasnoyarsk, Krasnoyarsk Krai
  - National Research Ogarev Mordovia State University ( Site 2648), Saransk, Mordoviya, Respublika
  - FSBI National Medical Oncology Research Center n.a. N.N. Blokhina ( Site 2634), Moscow, Moscow
  - Moscow Research Oncology Institute named after P.A. Hertsen ( Site 2631), Moscow, Moscow
  - Nizhegorodsky Regional Oncology Dispensary-chemotherapy department (Branch№1) ( Site 2639), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Samara Regional Clinical Oncology Center-Chemotherapy Dapartment ( Site 2649), Samara, Samara Oblast
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 2636), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 2646), Kazan', Tatarstan, Respublika
  - Tomsk Scientific Research Institute of Oncology-Chemotherapy ( Site 2638), Tomsk, Tomsk Oblast
  - Yaroslavl Regional SBIH Clinical Oncology Hospital ( Site 2641), Yaroslavl, Yaroslavl Oblast
- South Korea (5):
  - National Cancer Center ( Site 4065), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 4063), Seongnam-si, Kyonggi-do
  - Severance Hospital Yonsei University Health System ( Site 4062), Seoul
  - Asan Medical Center ( Site 4061), Seoul
  - Samsung Medical Center ( Site 4064), Seoul
- Spain (7):
  - Hospital Josep Trueta ( Site 2184), Girona, Gerona
  - Clinica Universitaria de Navarra ( Site 2181), Madrid, Madrid, Comunidad de
  - Hospital Vall D Hebron ( Site 2182), Barcelona
  - Hospital Clinic i Provincial ( Site 2185), Barcelona
  - Hospital Universitario Reina Sofia ( Site 2183), Córdoba
  - Hospital Clinico San Carlos ( Site 2187), Madrid
  - Hospital Universitario La Paz ( Site 2186), Madrid
- Sweden (3):
  - Karolinska Universitetssjukhuset Solna ( Site 2220), Solna, Stockholm County
  - Blod-och Tumorsjukdomar ( Site 2221), Uppsala, Uppsala County
  - Universitetssjukhuset i Linkoping. ( Site 2222), Linköping, Östergötland County
- Taiwan (5):
  - Changhua Christian Hospital ( Site 4095), Changhua
  - Taichung Veterans General Hospital ( Site 4094), Taichung
  - MacKay Memorial Hospital ( Site 4092), Taipei
  - Taipei Veterans General Hospital ( Site 4093), Taipei
  - Linkou Chang Gung Memorial Hospital ( Site 4091), Taoyuan District
- Turkey (Türkiye) (7):
  - Baskent Adana Dr Turgut Noyan Uygulama ve Arastirma Merkezi ( Site 2355), Adana
  - Cukurova Uni. Tip Fakultesi ( Site 2353), Adana
  - Baskent Universitesi Ankara Hastanesi ( Site 2354), Ankara
  - Ankara Universitesi Tıp Fakultesi Hastanesi ( Site 2350), Ankara
  - Medipol Universite Hastanesi ( Site 2352), Istanbul
  - Ege University Medical Faculty ( Site 2351), Izmir
  - I.E.U. Medical Point Hastanesi ( Site 2356), Izmir
- Ukraine (7):
  - Chernihiv Medical Center of Modern Oncology ( Site 2368), Chernihiv, Chernihiv Oblast
  - Municipal Enterprise "Bukovinian сlinical oncology сenter" ( Site 2366), Chernivtsi, Chernivetska Oblast
  - SO Grigoriev Institute for Medical Radiology and Oncology of NAMS of Ukraine ( Site 2363), Kharkiv, Kharkivs’ka Oblast’
  - MNE "Khmelnytskyi regional antitumor center" ( Site 2365), Khmelnitskyi, Khmelnytskyi Oblast
  - LISOD - Israeli Oncological Hospital MedX-ray International Group, LLC ( Site 2364), Kiev, Kyivska Oblast
  - Lviv State Regional Oncological Center ( Site 2361), Lviv, Lviv Oblast
  - The Municipal Enterprise Volyn Regional Medical Oncology Centre ( Site 2362), Lutsk, Volyn Oblast
- United Kingdom (8):
  - Bristol Haematology and Oncology Centre ( Site 2244), Bristol, Bristol, City of
  - Castle Hill Hospital-Academic Oncology ( Site 2252), Cottingham, East Riding Of Yorkshire
  - Beatson West of Scotland Cancer Centre ( Site 2247), Glasgow, Glasgow City
  - UCLH NHS Foundation Trust ( Site 2242), London, London, City of
  - Royal Marsden NHS Foundation Trust ( Site 2248), London, London, City of
  - Royal Marsden Hospital Sutton-Surrey ( Site 2241), Sutton, London, City of
  - Leicester Royal Infirmary. Univ. Hosp. of Leicester NHS Trust ( Site 2249), Leicester
  - The Christie Hospital NHS Foundation Trust ( Site 2243), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Van Gorp T, Cibula D, Lv W, Backes F, Ortac F, Hasegawa K, Lindemann K, Savarese A, Laenen A, Kim YM, Bodnar L, Barretina-Ginesta MP, Gilbert L, Pothuri B, Chen X, Flores MB, Levy T, Colombo N, Papadimitriou C, Buchanan T, Hanker LC, Eminowicz G, Rob L, Black D, Lichfield J, Lin G, Orlowski R, Keefe S, Lortholary A, Slomovitz B; ENGOT-en11/GOG-3053/KEYNOTE-B21 investigators. ENGOT-en11/GOG-3053/KEYNOTE-B21: a randomised, double-blind, phase III study of pembrolizumab or placebo plus adjuvant chemotherapy with or without radiotherapy in patients with newly diagnosed, high-risk endometrial cancer. Ann Oncol. 2024 Nov;35(11):968-980. doi: 10.1016/j.annonc.2024.08.2242. Epub 2024 Sep 14. PMID 39284383
- [Result] Slomovitz BM, Cibula D, Lv W, Ortac F, Hietanen S, Backes F, Kikuchi A, Lorusso D, Danska-Bidzinska A, Samouelian V, Barretina-Ginesta MP, Vulsteke C, Lai CH, Pothuri B, Zhang Y, Magallanes-Maciel M, Amit A, Guarneri V, Zagouri F, Bell M, Welz J, Eminowicz G, Hruda M, Willmott LJ, Lichfield J, Wang W, Orlowski R, Aktan G, Gladieff L, Van Gorp T. Pembrolizumab or Placebo Plus Adjuvant Chemotherapy With or Without Radiotherapy for Newly Diagnosed, High-Risk Endometrial Cancer: Results in Mismatch Repair-Deficient Tumors. J Clin Oncol. 2025 Jan 20;43(3):251-259. doi: 10.1200/JCO-24-01887. Epub 2024 Oct 16. PMID 39411812
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26257&tenant=MT_MSD_9011